CLINICAL TRIAL: NCT05407792
Title: Efficacy and Safety of Long-term Oral Administration of Staphylococcus Albicans Tablets in Patients With Acute Exacerbation and Stable Bronchiectasis: a Multicenter, Prospective Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Long-term Oral Staphylococcus Albicans Tablets in Patients With Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Principal Investigator, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-5-26-QFS
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral staphylococcus albicans tablet group.
  Interventions: Drug: Staphylococcus and Neisseria Tablets
- Control group (Other): On-demand treatment group
  Interventions: Other: On-demand treatment

INTERVENTIONS:
Drug: Staphylococcus and Neisseria Tablets — 0.3 mg/ tablet, 4 tablets each time, 3 times a day (Shandong Qilu Pharmaceutical Co., LTD.), the course of treatment was more than 3 months.
  Other Names: H37023540
  Arms: Experimental group
Other: On-demand treatment — At the time of enrollment, patients with acute exacerbation of bronchiectasis were given routine treatment. For patients with stable bronchiectasis at the time of enrollment, they are treated as needed (that is, according to the needs of the disease, receive corresponding treatment).
  Arms: Control group

SUMMARY:
The main purpose of this study is to investigate whether long-term oral administration of Staphylococcus albicans tablets can significantly reduce the number of acute exacerbations in patients with bronchiectasis. Secondary objective is to explore whether long-term oral administration of Staphylococcus albicans tablets can reduce the risk of hospitalization in patients with bronchiectasis and whether it can improve the quality of life of patients. Other purpose is to explore the regulatory effect of long-term oral administration of Staphylococcus albicans tablets on the immune function of patients with bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic airway purulent disease. The four factors of "vicious circle" play an important role in the occurrence, development and prognosis of bronchiectasis. Attempts to breaks the vicious circle may be beneficial to reduce the acute exacerbation of bronchiectasis. The main ingredients of Staphylococcus albicans tablets are the inactivated cells of Staphylococcus albus, Catarella catarrhalis and Bacillus subtilis. It may be beneficial to improve the non-specific immunity of patients and the specific immune function of respiratory mucosa, and reduce airway mucus secretion and secretion retention. There is not yet sufficient clinical evidence to support the immune function regulation and related efficacy of patients. Therefore, the efficacy of long-term oral administration of Staphylococcus albicans tablets in patients with bronchiectasis needs to be further confirmed by clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bronchiectasis diagnosed by clinical manifestations and chest HRCT according to the diagnostic criteria for bronchiectasis;

  * Patients with idiopathic or post-infectious bronchiectasis;

    * 18years old;

      * Patients should have at least 2 acute exacerbations within 1 year before enrollment;

        * Patients in either acute exacerbation or stable period can be included.

Exclusion Criteria:

* Cystic fibrosis;

  * Immunodeficiency, allergic bronchopulmonary aspergillosis, etc.;

    * Traction bronchiectasis caused by severe emphysema or advanced pulmonary fibrosis;

      * Still smoking;

        * Complicated with asthma or chronic obstructive disease Lung;

          * Patients with severe cardiovascular disease, severe neurological disease, or severe liver or kidney damage;

            * Malignant tumors;

              * Allergy to Staphylococcus albicans tablets;

                * Patients with a history of gastric ulcer or intestinal malabsorption;

                  * Pregnant or lactating women;

                    * patients with poor compliance;

                      * previous (within 6 months before the start of the study) or concurrently taking immunostimulating drugs (including thymosin, interferon, transfer factor, BCG, pneumonia vaccine and any kind of bacteria Extracts, such as Biostim, except for influenza vaccine) or immunosuppressants;

                        * Patients who are participating in or have participated in interventional clinical trials within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbations | Up to 12 months
Time to first exacerbation | Up to 12 months
Rate of readmission at 12 months | Up to 12 months
Number of acute exacerbations | up to 6 months
Number of acute exacerbations | Up to 3 months

SECONDARY OUTCOMES:
Change from Baseline Life Quality Score at 12 months | Up to 12 months
Change from Baseline FEV1 at 12 months | Up to 12 months
Change from Baseline FEV1/FVC at 12 months | Up to 12 months
Change from Baseline FEV1 % predicted at 12 months | Up to 12 months
Change from Baseline sputum volume at 12 months | Up to 12 months
Change from Baseline percentage of patients with yellow purulent sputum at 12 months | Up to 12 months
Change from Baseline percentage of patients with immune dysfunction at 12 months | Up to 12 months
Change from Baseline of percentage of patients with positive sputum culture | Up to 12 months
Number of Participants with adverse reactions | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China